CLINICAL TRIAL: NCT02581215
Title: Phase II Randomized, Double-Blind Study of mFOLFIRINOX Plus Ramucirumab Versus mFOLFIRINOX Plus Placebo in Advanced Pancreatic Cancer Patients: Hoosier Cancer Research Network GI14-198
Brief Title: Phase II Randomized Trial of mFOLFIRINOX +/- Ramucirumab in Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Walid Shaib, MD (Other)
Collaborators: Eli Lilly and Company (Industry); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor-Investigator, Walid Shaib, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCRN GI14-198
Record Dates: First submitted 2015-10-19; First posted 2015-10-20 (Estimated); Results first posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Cancer
Keywords: mFOLFIRINOX; Ramucirumab
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Ramucirumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Site pharmacy staff will be unblinded to the study treatment. Subjects, site investigators, site analysis teams, and other site personnel will be blinded to the study treatment.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Experimental Arm (Experimental): mFOLFIRINOX will be administered every 2 weeks, and consist of:
  * Oxaliplatin 85 mg/m2 over 2-4 hours
  * Irinotecan 165 mg/m2 over 90 minutes
  * 5-FU 2,400 mg/m2 as a 46-hour continuous infusion without the 5-FU bolus to decrease the risk of neutropenia.
  * Arm A will receive ramucirumab administered as an intravenous infusion over 60 minutes (infusion rate should not exceed 25 mg/min), at a fixed dose of 8 mg/kg every 2 weeks.
  Interventions: Drug: mFOLFIRINOX; Drug: Ramucirumab
- Arm B: Placebo Arm (Placebo Comparator): mFOLFIRINOX will be administered every 2 weeks, and consist of:
  * Oxaliplatin 85 mg/m2 over 2-4 hours
  * Irinotecan 165 mg/m2 over 90 minutes
  * 5-FU 2,400 mg/m2 as a 46-hour continuous infusion without the 5-FU bolus to decrease the risk of neutropenia.
  * Arm B will receive a placebo infusion every 2 weeks. Due to the double-blinded nature of this study, the volume of placebo will be calculated as if it were ramucirumab
  Interventions: Drug: mFOLFIRINOX; Other: Placebo

INTERVENTIONS:
Drug: mFOLFIRINOX — mFOLFIRINOX:
  * Oxaliplatin 85 mg/m2 over 2-4 hours
  * Irinotecan 165 mg/m2 over 90 minutes
  * 5-FU 2,400 mg/m2 as a 46-hour continuous infusion without the 5-FU bolus to decrease the risk of neutropenia.
Drug: Ramucirumab — Ramucirumab administered as an intravenous infusion over 60 minutes (infusion rate should not exceed 25 mg/min), at a fixed dose of 8 mg/kg every 2 weeks.
  Other Names: Cyramza
  Arms: Arm A: Experimental Arm
Other: Placebo — Placebo infusion with volume calculated as if it were ramucirumab every 2 weeks.
  Arms: Arm B: Placebo Arm

SUMMARY:
This is a phase II, multicenter, double-blinded, randomized, 2-arm trial evaluating the efficacy and safety of mFOLFIRINOX plus ramucirumab (Arm A) vs. mFOLFIRINOX plus placebo (Arm B) in 94 subjects with advanced pancreatic cancer, not amenable to curative treatment. Both arms will continue treatment until disease progression or unacceptable toxicity.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

EXPERIMENTAL ARM A:

* Oxaliplatin 85 mg/m^2 over 2-4 hours
* Irinotecan 165 mg/m^2 over 90 minutes
* 5-FU 2,400 mg/m^2 as a 46-hour continuous infusion without the 5-FU bolus to decrease the risk of neutropenia.
* Arm A will receive ramucirumab (RAM) administered as an intravenous infusion over 60 minutes (infusion rate should not exceed 25 mg/min), at a fixed dose of 8 mg/kg every 2 weeks.

CONTROL ARM B :

* Oxaliplatin 85 mg/m2 over 2-4 hours
* Irinotecan 165 mg/m2 over 90 minutes
* 5-FU 2,400 mg/m2 as a 46-hour continuous infusion without the 5-FU bolus to decrease the risk of neutropenia.
* Arm B will receive a placebo infusion every 2 weeks. Due to the double-blinded nature of this study, the volume of placebo will be calculated as if it were RAM.

In order to demonstrate adequate organ function, all screening labs must be obtained within 7 days prior to registration:

Hematological:

* Hemoglobin ≥ 9 g/dL
* Absolute Neutrophil Count (ANC) ≥ 1,500/mm^3
* Platelet Count (PLT) ≥ 100,000/mm^3

Renal:

* Creatinine ≤ 1.5 mg/dL or Creatinine clearance^1 ≥ 40 mL/min
* Albumin ≥ 2.5 g/dL

Hepatic:

* Bilirubin ≤ 1.5 mg/dL
* Aspartate aminotransferase (AST) ≤ 3 × ULN or < 5 xULN in the setting of liver metastases
* Alanine aminotransferase (ALT) ≤ 3 × ULN or < 5 xULN in the setting of liver metastases

Coagulation:

* International Normalized Ratio (INR) (Patients receiving warfarin must be switched to low molecular weight heparin and have achieved stable coagulation profile prior to first dose of protocol therapy) ≤1.5 and a partial thromboplastin time (PTT) (PTT/aPTT) < 1.5 x ULN

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information. .
* Age ≥ 18 years at the time of consent.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1 within 7 days prior to registration.
* Histologic or cytological diagnosis of recurrent or metastatic pancreas adenocarcinoma (PCA) who present for first line chemotherapy treatment.
* No prior first line systemic treatment (prior adjuvant or neoadjuvant treatment is permitted). Subjects whose disease has progressed after 6 months of last systemic chemotherapy or chemo-radiation in the adjuvant or neoadjuvant setting are eligible.
* Measurable disease determined using guidelines of Response Evaluation Criteria In Solid Tumors (RECIST 1.1). Baseline tumor assessment should be performed using high resolution computed tomography (CT) scans or magnetic resonance imaging (MRI).
* Urine protein < 1+ on dipstick test or routine urinalysis. If the proteinuria on these tests is ≥2+, then a 24-hour urine test must be collected and must demonstrate < 1g proteins in 24 hours to allow participation.
* Estimated life expectancy of >12 weeks, as assessed by the site investigator.
* If sexually active, must be postmenopausal, surgically sterile, or using effective contraception (hormonal or barrier methods) due to unknown risk of teratogenicity of ramucirumab

Exclusion Criteria:

* Subjects with histology other than adenocarcinoma; Examples include: neuroendocrine tumors, acinar cell cancer, sarcoma or lymphoma of the pancreas.
* Ongoing or active infection.
* Symptomatic congestive heart failure, unstable angina pectoris, symptomatic or poorly controlled cardiac arrhythmia. Symptomatic heart failure per New York Heart Association (NYHA) Class II-IV.
* Uncontrolled or poorly-controlled hypertension (>160 mmHg systolic or > 100 mmHg diastolic for >4 weeks) despite standard medical management.
* Acute or sub-acute intestinal obstruction.
* Interstitial pneumonia or interstitial fibrosis of the lung, which in the opinion of the site investigator could compromise the subject or the study.
* Pleural effusion or ascites that causes > grade 1 dyspnea.
* Cirrhosis at a level of Child-Pugh B (or worse) or cirrhosis (any degree) with a history of hepatic encephalopathy or clinical meaningful ascites resulting from cirrhosis; clinically meaningful ascites is defined as ascites resulting from cirrhosis and requiring ongoing treatment with diuretics and/or paracentesis.
* Grade 3 or higher bleeding event ≤ 3 months prior to randomization.
* Experience of any arterial thrombotic or arterial thromboembolic events, including, but not limited to myocardial infarction, transient ischemic attack, or cerebrovascular accident, ≤ 6 months prior to randomization.
* History of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 3 months prior to randomization.
* Documented and/or symptomatic or known brain or leptomeningeal metastases.
* GI perforation/fistula
* Documented and/or symptomatic or known brain or leptomeningeal metastases.
* Severely immune-compromised (other than being on steroids), including known HIV infection.
* Concurrent active malignancy other than adequately treated non-melanoma skin cancer, other noninvasive carcinoma, or in situ neoplasm. A subject with previous history of malignancy is eligible, provided that he/she has been disease free for > 3 years.
* Breast-feeding or pregnant.
* Prior autologous or allogeneic organ or tissue transplantation.
* Known allergy to any of the treatment components.
* Major surgery within 28 days prior to the first dose of protocol therapy, or minor surgery/subcutaneous venous access device placement within 2 days prior to first dose of protocol therapy. The patient has elective or planned major surgery to be performed during the course of the clinical trial.
* Any condition that does not permit compliance with the study schedule including psychological, geographical or medical.
* Receiving medications that can effect clotting ability: warfarin, aspirin (once-daily aspirin use- maximum dose 325 mg/day is permitted), nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents. .
* Serious or non-healing wound, ulcer, or bone fracture within 28 days prior to first dose of protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-09-11 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2022-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walid Shaib, MD, Principal Investigator — Emory University
Locations (8):
- United States (8):
  - Mayo Clinic-Arizona, Scottsdale, Arizona
  - Emory University: Winship Cancer Institute, Atlanta, Georgia
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Community Healthcare System, Munster, Indiana
  - University of Louisville, James Graham Brown Cancer Center, Louisville, Kentucky
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Thomas Jefferson University Kimmel Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Shaib WL, Manali R, Liu Y, El-Rayes B, Loehrer P, O'Neil B, Cohen S, Khair T, Robin E, Huyck T, Bekaii-Saab T. Phase II randomised, double-blind study of mFOLFIRINOX plus ramucirumab versus mFOLFIRINOX plus placebo in advanced pancreatic cancer patients (HCRN GI14-198). Eur J Cancer. 2023 Aug;189:112847. doi: 10.1016/j.ejca.2023.02.030. Epub 2023 Mar 11. PMID 37268519
- See also: Hoosier Cancer Research Network Website — http://www.hoosiercancer.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Experimental Arm: mFOLFIRINOX will be administered every 2 weeks, and consist of:
  * Oxaliplatin 85 mg/m2 over 2-4 hours
  * Irinotecan 165 mg/m2 over 90 minutes
  * 5-FU 2,400 mg/m2 as a 46-hour continuous infusion without the 5-FU bolus to decrease the risk of neutropenia.
  * Arm A will receive ramucirumab administered as an intravenous infusion over 60 minutes (infusion rate should not exceed 25 mg/min), at a fixed dose of 8 mg/kg every 2 weeks.
  mFOLFIRINOX: mFOLFIRINOX:
  * Oxaliplatin 85 mg/m2 over 2-4 hours
  * Irinotecan 165 mg/m2 over 90 minutes
  * 5-FU 2,400 mg/m2 as a 46-hour continuous infusion without the 5-FU bolus to decrease the risk of neutropenia.
  Ramucirumab: Ramucirumab administered as an intravenous infusion over 60 minutes (infusion rate should not exceed 25 mg/min), at a fixed dose of 8 mg/kg every 2 weeks.
- Arm B: Placebo Arm: mFOLFIRINOX will be administered every 2 weeks, and consist of:
  * Oxaliplatin 85 mg/m2 over 2-4 hours
  * Irinotecan 165 mg/m2 over 90 minutes
  * 5-FU 2,400 mg/m2 as a 46-hour continuous infusion without the 5-FU bolus to decrease the risk of neutropenia.
  * Arm B will receive a placebo infusion every 2 weeks. Due to the double-blinded nature of this study, the volume of placebo will be calculated as if it were ramucirumab
  mFOLFIRINOX: mFOLFIRINOX:
  * Oxaliplatin 85 mg/m2 over 2-4 hours
  * Irinotecan 165 mg/m2 over 90 minutes
  * 5-FU 2,400 mg/m2 as a 46-hour continuous infusion without the 5-FU bolus to decrease the risk of neutropenia.
  Placebo: Placebo infusion with volume calculated as if it were ramucirumab every 2 weeks.
Period: Overall Study
Arm/Group | Arm A: Experimental Arm | Arm B: Placebo Arm
Started | 42 | 42
Completed | 42 | 40
Not Completed | 0 | 2
Not completed — Screen Failure Before Therapy Start | 0 | 1
Not completed — Eligibility Criteria Not Met | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Experimental Arm | Arm B: Placebo Arm | Total
Number analyzed (Participants) | 42 | 40 | 82
Age, Continuous [Median (Full Range); unit: years] | 62 [40 to 79] | 65 [44 to 77] | 63 [40 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 23 | 20 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 41 | 35 | 76
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 35 | 34 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 42 | 40 | 82

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) at 9 Month
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  PFS is defined as time of registration until disease progression met by RECIST 1.1 or death from any cause.
Time Frame: 9 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Experimental Arm | Arm B: Placebo Arm
Number analyzed (Participants) | 42 | 40
Percentage of participants | 25.1 [11.6 to 41.3] | 35 [19.8 to 50.6]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined by the date of randomization to date of death from any cause.
Time Frame: Up to a maximum of 53 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Experimental Arm | Arm B: Placebo Arm
Number analyzed (Participants) | 42 | 40
Months | 10.3 [6 to 11.8] | 9.7 [6.4 to 15.9]

3. Secondary Outcome: Response Rate (RR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  Overall Response (OR) = CR + PR.
Time Frame: Up to 44 months
Population: The analysis population for the endpoint Response Rate (RR) was defined as all participants with at least one post-baseline disease assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Experimental Arm | Arm B: Placebo Arm
Number analyzed (Participants) | 34 | 31
Percentage of participants | 17.7 | 22.6

4. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events will be assessed to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) version 4.
Time Frame: From date of first dose until 30 days after the last treatment, assessed up to 44 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Experimental Arm | Arm B: Placebo Arm
Number analyzed (Participants) | 42 | 40
Participants | 42 | 40

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored up to a maximum of 53 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored up to 44 months.
Arm/Group | Arm A: Experimental Arm | Arm B: Placebo Arm
All-Cause Mortality (participants affected / at risk) | 33/42 | 35/40
Serious Adverse Events (participants affected / at risk) | 19/42 | 17/40
Other Adverse Events (participants affected / at risk) | 41/42 | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Experimental Arm (N=42) | Arm B: Placebo Arm (N=40)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 2 (2)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 2 (2) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
CONFUSION (Psychiatric disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 3 (3) | 1 (3)
DUODENAL OBSTRUCTION (Gastrointestinal disorders) | 3 (3) | 0 (0)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
ESOPHAGITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 1 (2) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 1 (1) | 0 (0)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 1 (1) | 0 (0)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 1 (1) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (2) | 0 (0)
PAIN (General disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
SEPSIS (Infections and infestations) | 3 (6) | 3 (4)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 3 (3) | 2 (2)
BLADDER INFECTION (Infections and infestations) | 0 (0) | 1 (1)
COLONIC OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
DEATH NOS (General disorders) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
HEPATOBILIARY DISORDERS - OTHER, SPECIFY (Hepatobiliary disorders) | 0 (0) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
RENAL CALCULI (Renal and urinary disorders) | 0 (0) | 1 (1)
TRANSIENT ISCHEMIC ATTACKS (Nervous system disorders) | 0 (0) | 1 (1)
UPPER GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 2 (2)
VISCERAL ARTERIAL ISCHEMIA (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Experimental Arm (N=42) | Arm B: Placebo Arm (N=40)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 (2) | 0 (0)
ABDOMINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 20 (32) | 18 (28)
ABDOMINAL SOFT TISSUE NECROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 10 (19) | 6 (9)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 11 (23) | 10 (26)
ALLERGIC REACTION (Immune system disorders) | 3 (3) | 4 (5)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (10)
ANEMIA (Blood and lymphatic system disorders) | 14 (44) | 12 (46)
ANOREXIA (Metabolism and nutrition disorders) | 20 (33) | 16 (25)
ANXIETY (Psychiatric disorders) | 6 (6) | 9 (10)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 7 (15) | 5 (8)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 (8) | 7 (9)
BLOATING (Gastrointestinal disorders) | 1 (1) | 1 (1)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (Blood and lymphatic system disorders) | 3 (3) | 3 (7)
BLOOD BILIRUBIN INCREASED (Investigations) | 5 (12) | 3 (6)
BLURRED VISION (Eye disorders) | 1 (2) | 3 (3)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
CHILLS (General disorders) | 2 (4) | 3 (3)
COLITIS (Gastrointestinal disorders) | 1 (1) | 2 (2)
CONFUSION (Psychiatric disorders) | 2 (2) | 2 (2)
CONSTIPATION (Gastrointestinal disorders) | 11 (13) | 11 (16)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (5)
CREATININE INCREASED (Investigations) | 1 (1) | 1 (4)
DEHYDRATION (Metabolism and nutrition disorders) | 8 (9) | 8 (10)
DEPRESSION (Psychiatric disorders) | 8 (8) | 4 (4)
DIARRHEA (Gastrointestinal disorders) | 29 (58) | 27 (56)
DIZZINESS (Nervous system disorders) | 5 (5) | 3 (4)
DRY MOUTH (Gastrointestinal disorders) | 3 (3) | 1 (1)
DUODENAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSARTHRIA (Nervous system disorders) | 1 (1) | 1 (1)
DYSESTHESIA (Nervous system disorders) | 2 (2) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 7 (8) | 2 (2)
DYSPEPSIA (Gastrointestinal disorders) | 3 (3) | 2 (2)
DYSPHAGIA (Gastrointestinal disorders) | 2 (2) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (10)
EDEMA LIMBS (General disorders) | 6 (7) | 2 (2)
ENDOCRINE DISORDERS - OTHER, SPECIFY (Endocrine disorders) | 1 (1) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
ESOPHAGEAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
ESOPHAGITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 3 (4)
FATIGUE (General disorders) | 28 (66) | 25 (54)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
FEVER (General disorders) | 3 (3) | 7 (8)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
GAIT DISTURBANCE (General disorders) | 1 (1) | 0 (0)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 7 (7) | 8 (11)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 4 (5) | 2 (2)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 6 (9) | 3 (3)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (7)
GUM INFECTION (Infections and infestations) | 2 (3) | 0 (0)
HEADACHE (Nervous system disorders) | 6 (8) | 2 (8)
HEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 2 (2)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 8 (13) | 9 (23)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 (4) | 1 (1)
HYPERTENSION (Vascular disorders) | 12 (24) | 10 (24)
HYPERURICEMIA (Metabolism and nutrition disorders) | 3 (4) | 5 (5)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 7 (14) | 5 (14)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 5 (6) | 4 (9)
HYPOKALEMIA (Metabolism and nutrition disorders) | 13 (22) | 12 (31)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 8 (10) | 6 (11)
HYPONATREMIA (Metabolism and nutrition disorders) | 9 (13) | 4 (6)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (6)
HYPOTENSION (Vascular disorders) | 2 (3) | 4 (5)
HYPOTHYROIDISM (Endocrine disorders) | 4 (4) | 2 (2)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 2 (2) | 2 (2)
INFUSION RELATED REACTION (General disorders) | 3 (5) | 1 (1)
INSOMNIA (Psychiatric disorders) | 4 (4) | 5 (6)
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 1 (1) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
LYMPHEDEMA (Vascular disorders) | 1 (1) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 4 (16) | 2 (4)
LYMPHOCYTE COUNT INCREASED (Investigations) | 1 (1) | 0 (0)
MALABSORPTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
MUCOSAL INFECTION (Infections and infestations) | 2 (3) | 0 (0)
MUCOSITIS ORAL (Gastrointestinal disorders) | 6 (9) | 5 (6)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 29 (70) | 28 (51)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 3 (7) | 4 (7)
NEUTROPHIL COUNT DECREASED (Investigations) | 17 (35) | 14 (24)
NON-CARDIAC CHEST PAIN (General disorders) | 2 (2) | 1 (2)
ORAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
PAIN (General disorders) | 4 (4) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
PARESTHESIA (Nervous system disorders) | 4 (9) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 5 (7) | 4 (7)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 21 (33) | 21 (42)
PERITONEAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PHARYNGEAL MUCOSITIS (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 10 (45) | 13 (45)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 2 (5) | 4 (4)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL CALCULI (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 1 (4) | 0 (0)
SALIVARY DUCT INFLAMMATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
SINUS PAIN (Nervous system disorders) | 1 (1) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1) | 4 (8)
SINUSITIS (Infections and infestations) | 2 (2) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
SOFT TISSUE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
THROMBOEMBOLIC EVENT (Vascular disorders) | 5 (6) | 7 (9)
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 1 (1) | 0 (0)
TREMOR (Nervous system disorders) | 1 (2) | 0 (0)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (1) | 2 (2)
URINARY FREQUENCY (Renal and urinary disorders) | 3 (3) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 4 (5) | 5 (6)
URINARY TRACT PAIN (Renal and urinary disorders) | 2 (2) | 0 (0)
VOMITING (Gastrointestinal disorders) | 23 (39) | 15 (37)
WATERING EYES (Eye disorders) | 1 (1) | 0 (0)
WEIGHT GAIN (Investigations) | 1 (2) | 3 (3)
WEIGHT LOSS (Investigations) | 25 (30) | 18 (20)
WHITE BLOOD CELL DECREASED (Investigations) | 8 (22) | 5 (21)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (1)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BLADDER INFECTION (Infections and infestations) | 0 (0) | 1 (1)
BRONCHIAL INFECTION (Infections and infestations) | 0 (0) | 1 (2)
BRUISING (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CARDIAC DISORDERS - OTHER, SPECIFY (Cardiac disorders) | 0 (0) | 1 (1)
CATHETER RELATED INFECTION (Infections and infestations) | 0 (0) | 1 (1)
CONJUNCTIVITIS (Eye disorders) | 0 (0) | 1 (1)
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 0 (0) | 1 (2)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
EAR AND LABYRINTH DISORDERS - OTHER, SPECIFY (Ear and labyrinth disorders) | 0 (0) | 1 (2)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 1 (1)
EDEMA TRUNK (General disorders) | 0 (0) | 1 (1)
ESOPHAGEAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
FACIAL MUSCLE WEAKNESS (Nervous system disorders) | 0 (0) | 1 (1)
FECAL INCONTINENCE (Gastrointestinal disorders) | 0 (0) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 3 (3)
FLU LIKE SYMPTOMS (General disorders) | 0 (0) | 1 (1)
FLUSHING (Vascular disorders) | 0 (0) | 1 (1)
HEARING IMPAIRED (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEMATOMA (Vascular disorders) | 0 (0) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 0 (0) | 2 (2)
HEPATOBILIARY DISORDERS - OTHER, SPECIFY (Hepatobiliary disorders) | 0 (0) | 1 (1)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
IMMUNE SYSTEM DISORDERS - OTHER, SPECIFY (Immune system disorders) | 0 (0) | 1 (1)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INR INCREASED (Investigations) | 0 (0) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
NEURALGIA (Nervous system disorders) | 0 (0) | 1 (1)
ORAL DYSESTHESIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 1 (1)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PANCREATIC ENZYMES DECREASED (Investigations) | 0 (0) | 1 (1)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
STOMACH PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
SURGICAL AND MEDICAL PROCEDURES - OTHER, SPECIFY (Surgical and medical procedures) | 0 (0) | 1 (1)
URINE DISCOLORATION (Renal and urinary disorders) | 0 (0) | 1 (1)
VASCULAR DISORDERS - OTHER, SPECIFY (Vascular disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/15/NCT02581215/Prot_SAP_000.pdf